CLINICAL TRIAL: NCT06904690
Title: JACARDI: A eHealth and Health Literacy Educational Training to Support Older Patients With Type II Diabetes
Acronym: JACARDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INRCA_003_2025
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; eHealth literacy; elderly subjects; wellbeing; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Training Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diabetic subjects (Experimental): Subjects with type 2 diabetes who have low eHealth literacy.
  Interventions: Other: Educational training

INTERVENTIONS:
Other: Educational training — The educational training is divided into the following five modules:
  Module 1: Raising Awareness of eHealth and Health Literacy (Introduction to the aims and context of JACARDI and diabetes);
  Module 2: Acquiring New Knowledge (Health Literacy and Self-Management of Diabetes);
  Module 3: Acquiring New Knowledge (Technological and Non-Technological Strategies to Support the Self-Management of Diabetes);
  Module 4: Practicing New Skills (Usability with Practice Sessions);
  Module 5: Self-Evaluation and Sustainability of Improvement (Final Questionnaire).
  The training will be conducted over 10 weeks (one session every other week), with each session lasting an average of 90 minutes.

SUMMARY:
The JACARDI trial is a multicenter study involving an educational training, with the general objective to improve the eHealth of older adults in relation to the management of type 2 diabetes.

DETAILED DESCRIPTION:
The JACARDI trial is a multicentric study organized as a blended didactic and interactive educational training, with the general objective to improve the eHealth of older adults in relation to the management of type 2 diabetes, thus contributing to independent living, and reduce risks of negative consequences for the health status and quality of life.

The trial will be preceded by a pre-study, needed to personalize and finalize the contents of the training, together with the beneficiaries of the study. In particular, during the pre-study, a population with similar characteristics of the target group will be involved in focus groups to refine the contents and practicalities of the training before the recruitment starts.

The primary end-point of the JACARDI trial is the improvement of the eHealth literacy after the conduction of the training, to be measured through the eHEALS scale, after 10 weeks of training. The training consisting of 5 modules and will be conducted over 10 weeks (one session every other week), with each session lasting an average of 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Low eHealth literacy (eHeals scale ≤ 29)
* No acute or untreated medical problems
* Mini Mental State Examination (MMSE) ≥ 24
* Geriatric Depression Scale (GDS) < 2

Exclusion Criteria:

* A myocardial infarction or stroke within 6 months
* Painful arthritis, spinal stenosis, amputation, painful foot lesions or neuropathy limiting balance and mobility
* Uncontrolled hypertension
* Advanced Parkinson's disease or other neuromuscular disorder
* Metastatic cancer or immunosuppressive therapy
* Significant visual or hearing impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
eHealth literacy | Baseline and 10, 14 and 34 weeks later
  Measured using the eHealth Literacy Scale (eHEALS). Scores range from 8 to 40, with higher scores indicating higher eHealth literacy.

SECONDARY OUTCOMES:
Health literacy | Baseline and 10, 14 and 34 weeks later
  Measured using the 16 items European Health Literacy Survey Questionnaire (HLS-EU-Q16). Each of the 16 items is answered by choosing one response from those available: 'very difficult', 'fairly difficult', 'fairly easy' and 'very easy. The four response categories are binarized (1 = "very easy / "fairly easy"; 0 = "very difficult" / "fairly difficult") and added together to form a total score: "adequate" (13-16 points), "problematic" (9-12 points) and "inadequate" (1-8 points).
Health-related quality of life | Baseline and 10, 14 and 34 weeks later
  Measured using the 5-level EQ-5D version (EQ-5D-5L) from the EuroQol Group. It includes one item addressing each of five dimensions (mobility, self-care, usual activity, pain/discomfort, and anxiety/depression). Participants rate each of these items from 1 of the 5 levels: no problems, slight problems, moderate problems, severe problems, or unable to/extreme. A composite health state is then defined by combining the levels for each dimension into a 5-digit number.
Psychological well-being | Baseline and 10, 14 and 34 weeks later
  Measured by the Psychological Wellbeing Scale (PWB). A self-administered questionnaire consisting of 18 items that investigates the degree of psychological well-being by exploring six dimensions: self-acceptance, positive relationships with others, autonomy, environmental control, personal growth, and purpose of life. The questionnaire consists of 18 items on a 4-step Likert scale. The higher numbers indicate greater agreement with positive statements or disagreement with negative statements. Scores are calculated for each of the six dimensions by summing or averaging the responses to the items within that dimension.
Diabetes related emotional distress | Baseline and 10, 14 and 34 weeks later
  Measured by the Problem Areas in Diabetes Questionnaire (PAID). The PAID is a self-report questionnaire that contains 20 items describing negative emotions related to diabetes (e.g. fear, anger, frustration) commonly experienced by patients with diabetes. Each question has five possible answers with a value from 0 ("no problem") to 4 ("a serious problem").Scores range from 0 - 100, higer scores indicate worse outcome.
Health-related quality of life | Baseline and 10, 14 and 34 weeks later
  Measured using the EQ visual analogue scale (EQ VAS) of the 5-level EQ-5D version (EQ-5D-5L) from the EuroQol Group. It measures self-rated health status utilizing a vertically oriented visual analogue scale where 100 represents the "best imaginable health state" and 0 represents the "worst imaginable health state." Respondents are asked to rate their current health by placing a mark along this continuum. The VAS provides a quantitative measure of the patient's perceived health state.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Bevilacqua, Principal Investigator — IRCCS INRCA, Ancona, Italy
Locations (2):
- Italy (2):
  - AOU Ospedaliera Marche, Ancona
  - IRCCS INRCA Hospital, Ancona

IPD SHARING:
Plan to Share IPD: No